CLINICAL TRIAL: NCT02518932
Title: The Effect of VTC-G15 (a Pentapeptide Cleavage Product og GLP-1) on Whole Body Glucose Metabolism in Man
Acronym: LVKGR
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elahi, Dariush, PhD (Individual)
Collaborators: ICON plc (Industry); Massachusetts General Hospital (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: VTC-G15
Record Dates: First submitted 2015-06-25; First posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug GLP-1 (32-36) Amide (Experimental): To examine insulinomemtic of the last 5 amino acids of GLP-1 from 60-180 min during a 4 hour hyperglycemic clamp
  Interventions: Drug: Last 5 amino acids of GLP-1
- Placebo (Placebo Comparator): To examine the effect of saline on glucose uptake
  Interventions: Drug: placebo saline

INTERVENTIONS:
Drug: Last 5 amino acids of GLP-1 — To examine insulinomimetic properties of LVKGR
  Other Names: VTC-G15; LVKGR
  Arms: Drug GLP-1 (32-36) Amide
Drug: placebo saline
  Arms: Placebo

SUMMARY:
To asses the modulating properties of the cleaved pentapeptide product of GLP-1 amide.

DETAILED DESCRIPTION:
The investigators have previously demonstrated that infusion of the pentapeptide during hyperglycemic clamps in dogs significantly increases the glucose infusion rate necessary to maintain stable hyperglycemia without any significant differences in insulin or glucagon secretion. The present study's aim is to examine whether this also occurs in humans. It may be necessary to examine a dose response curve. Specifically, in twenty healthy volunteers glucose infusion rate during the peptide infusion will be compared to the glucose infusion rate during saline administration during a 4 hour hyperglycemic clamp, in a cross over design(mg/kg/min).

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-25;
* 33-38

Exclusion Criteria:

* T2D
* T1D
* Hypoglycemic agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The effect of VTC-G15 on whole body glucose metabolism in man will be assessed by comparison of amont of glucose infusion during the peptide infusion compared to amount of infusion during placebo infusion (saline) mg/kg/min. | one year

SECONDARY OUTCOMES:
THe effect of VTC-G15(A pentapeptide cleavage product of GLP-1) on whole body glucose metabolism in man. | one year
  changes in insulin or glucagon release.

CONTACTS AND LOCATIONS:
Overall Officials: Dariush Elahi, PhD, Principal Investigator — ICON plc, 8307 Gault Lane, San Antonio TX 78209
Locations (1):
- ICON PLC, San Antonio, Texas, United States